CLINICAL TRIAL: NCT05715866
Title: Effect of Non-invasive Stimulation Through Nesa and Therapeutic Exercise on Sleep Disturbances on Alzheimer's Disease Patients. Randomized Multicenter Clinical Trial
Brief Title: Non-invasive Stimulation Through Nesa and Therapeutic Exercise on Sleep Disturbances on Alzheimer's Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Esther del Carmen Teruel Hernández, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ET_2021
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; sleep disorders
MeSH Terms: conditions — Alzheimer Disease; Sleep Wake Disorders | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Random intervention model
Who Masked: Outcomes Assessor
Masking Description: The evaluators of all the results and the main caregivers of the participating patients will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-invasive neurostimulation experimental group (NEG) (Experimental): The non-invasive neuromodulation experimental group, made up of 10 participants, are treated 20 sessions with the NXSignal non-invasive neuromodulation device (NESA)
  Interventions: Device: non-invasive neuromodulation through the Nesa device
- Experimental group Therapeutic Exercise (TEG) (Experimental): The experimental group of therapeutic exercise, made up of 10 participants, receives 3 weekly sessions of one hour duration for 16 weeks, and 1 weekly session until week 20, of an adapted program of cardiovascular exercises in a small group format, supervised by a physical therapist.
  Interventions: Procedure: therapeutic exercise
- Control group (CG) (Sham Comparator): The control group, made up of 10 participants, the caregivers receive recommendations about sleep habits through an information brochure.
  Interventions: Behavioral: sleep hygiene measures

INTERVENTIONS:
Device: non-invasive neuromodulation through the Nesa device — patients receive non-invasive neurostimulation through the Nesa device
  Arms: non-invasive neurostimulation experimental group (NEG)
Procedure: therapeutic exercise — patients receive adapted therapeutic exercise
  Arms: Experimental group Therapeutic Exercise (TEG)
Behavioral: sleep hygiene measures — caregivers receive a brochure with sleep hygiene measures
  Arms: Control group (CG)

SUMMARY:
The purpose of this study is to know the effectiveness of an adapted therapeutic exercise program and its comparison with non-invasive neuromodulation through the NESA device, and both treatments with a control group, to improve sleep disturbances and cognitive function in patients with dementia, and improves the quality of life of their caregivers.

DETAILED DESCRIPTION:
Sleep disorders affect 30% of patients with dementia, being a very frequent symptom and appearing above all in the more advanced phases, and contribute to the risk of greater institutionalization, overload, and poorer quality of life for caregivers and abuse of sleep psychoactive drugs. Sleep disturbance is frequent in dementia, appearing especially in the more advanced stages. Non-pharmacological treatments are emerging as procedures of first choice to improve night rest in patients with Alzheimer's disease, however, given that the drugs do not remove the amyloid deposits that are formed or prevent their formation, and they have side effects adverse effects, the need arises to look for other options to improve the functioning of neuronal plasticity.

In Alzheimer's disease, therapeutic exercise has preventive and delayed effects against cognitive deterioration, in addition, it has been associated with changes in the circadian rhythm phases, however, there are no published controlled studies that analyze the isolated effects of exercise on sleep disturbances in patients with dementia.

Likewise, non-invasive neuromodulation through the NESA device consists of an alteration of the nervous activity through the delivery of microcurrents, which leads to a series of neuromodulated responses of the ANS neural cascades that gives rise to variations in the responses. endogenous of those dysfunctional or pathological bioelectrical systems.

Stimulation of the pineal gland through its sympathetic innervation results in the production of melatonin, a synchronizer of the circadian rhythm. In dementia there is a decrease in the level of melatonin, with non-invasive neuromodulation the pineal gland could be stimulated through its sympathetic innervation, resulting in the production of melatonin.

Objective: To know the effectiveness of an adapted therapeutic exercise program and its comparison with non-invasive neuromodulation through the NESA device, and both treatments with a control group, to improve sleep disturbances and cognitive function in patients with dementia. and improves the quality of life of their caregivers.

Methodology: This is a multicenter randomized clinical trial, with 30 patients diagnosed with dementia from two associations in the Region of Murcia for patients with Alzheimer's disease and other dementias, divided into three treatment groups, one of whom will receive non-invasive neuromodulation through NESA, another will be treated with therapeutic exercise, and a third control group, whose relatives will be given a brochure with sleep hygiene measures at the beginning of the study. The treatment will last 2 months for the neuromodulation group and 5 months for the therapeutic exercise group.

The measurements of the results are made individually, and under the same conditions for all the patients. These focus on cognitive and sleep variables for the patient with dementia and psychosocial variables to measure the quality of life of the caregiver. Each patient will be evaluated in four moments:

1. The first assessment before beginning the intervention period (pre-treatment)
2. The second evaluation in the middle of the treatment.
3. The third assessment at the end of the intervention period. (post-treatment)
4. The fourth two months after finishing the intervention. (tracing) The evaluators are masked. To measure the sleep variable, we have used various scales that reveal data on quality, efficiency, and quantity: Pittsburg sleep quality index (PSQI) and test de Epworth. To measure the cognitive variable for the patient with dementia, a scale has been used: Mini-Cognitive Exam Test (MEC). To measure the quality-of-life variable for the caregiver of the patient with dementia, the following scales have been used: Zarit scale and visual analogue scale (EVA).

ELIGIBILITY:
Inclusion Criteria:

* obtaining a medical diagnosis of dementia equal to or greater than mild according to the Reisberg Global Deterioration Scale (GDS)
* having stable medical and pharmacological conditions, as well as their ability to perform physical activity and follow instructions verbal

Exclusion Criteria:

* wearing a pacemaker
* presenting internal bleeding
* skin with ulcerations
* acute febrile processes
* diagnosis of cancer
* phobia of electricity
* comorbidity that affects the sleep

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality | [Time frame: Measurement of change: before treatment (baseline), at two months (mid-treatment), at five months (end of treatment), and at 7 months of treatment (follow-up period)
  We want to see if there are improvements in the quality, efficiency, and quantity of sleep. The Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale (ESS) will be combined to report changes in the patient's sleep quality.
Change in cognitive status | [Time frame: Measurement of change: before treatment (baseline), at two months (mid-treatment), at five months (end of treatment), and at 7 months of treatment (follow-up period)
  we want to see the cognitive improvement through the Mini-Cognitive Test (Mini-Cognitive Test. Lobo et al. Spanish version of the Mini Examination of the Mental State)
Change in quality of life | [Time frame: Measurement of change: before treatment (baseline), at two months (mid-treatment), at five months (end of treatment), and at 7 months of treatment (follow-up period)
  We want to see if the quality of life of caregivers of patients with dementia improves when their relatives receive treatment. The visual analogue scale (EVA) and the caregiver burden scale (Zarit) will be combined to report changes in the caregiver's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Esther del Carmen Teruel Hernández, MsC, Principal Investigator — Universidad de Murcia; Antonia Gomez-Conesa., Ph. D., Study Director — Universidad de Murcia; Jose A. Lopez Pina, Ph.D., Study Director — Universidad de Murcia; Sonia Souto Camba, Ph.D., Study Director — Universidade da Coruña
Locations (2):
- Spain (2):
  - AFADE: Association of relatives of Alzheimer's and other dementias, Alcantarilla, Murcia
  - AFAMUR, Association of relatives of Alzheimer's patients, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teruel-Hernandez E, Lopez-Pina JA, Souto-Camba S, Baez-Suarez A, Medina-Ramirez R, Gomez-Conesa A. Improving Sleep Quality, Daytime Sleepiness, and Cognitive Function in Patients with Dementia by Therapeutic Exercise and NESA Neuromodulation: A Multicenter Clinical Trial. Int J Environ Res Public Health. 2023 Nov 6;20(21):7027. doi: 10.3390/ijerph20217027. PMID 37947583